CLINICAL TRIAL: NCT02641444
Title: Antiretroviral Localization in Gut-Associated Lymphoid Tissue and Lower Female Genital Tract Tissue of HIV+ Subjects
Status: Terminated | Type: Observational
Why Stopped: Study team finished their analysis.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Angela Kashuba, PharmD, Professor, Division of Pharmacotherapy and Experimental Therapeutics, Eshelman School of Pharmacy, University of North Carolina, Chapel Hill
Other Study IDs: 15-2865
Record Dates: First submitted 2015-12-17; First posted 2015-12-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-04

CONDITIONS: HIV
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Efavirenz: Receiving efavirenz as part of their HIV regimen. Will undergo blood plasma collection, cervical and vaginal biopsy, and colonoscopy with ileal and rectal biopsy.
  Interventions: Procedure: Blood plasma collection; Procedure: Cervical and Vaginal Biopsy; Procedure: Colonoscopy with Ileal and Rectal Biopsy
- Atazanavir: Receiving atazanavir as part of their HIV regimen. Will undergo blood plasma collection, cervical and vaginal biopsy, and colonoscopy with ileal and rectal biopsy.
  Interventions: Procedure: Blood plasma collection; Procedure: Cervical and Vaginal Biopsy; Procedure: Colonoscopy with Ileal and Rectal Biopsy
- Raltegravir: Receiving raltegravir as part of their HIV regimen. Will undergo blood plasma collection, cervical and vaginal biopsy, and colonoscopy with ileal and rectal biopsy.
  Interventions: Procedure: Blood plasma collection; Procedure: Cervical and Vaginal Biopsy; Procedure: Colonoscopy with Ileal and Rectal Biopsy
- Maraviroc: Receiving maraviroc as part of their HIV regimen. Will undergo blood plasma collection, cervical and vaginal biopsy, and colonoscopy with ileal and rectal biopsy.
  Interventions: Procedure: Blood plasma collection; Procedure: Cervical and Vaginal Biopsy; Procedure: Colonoscopy with Ileal and Rectal Biopsy

INTERVENTIONS:
Procedure: Blood plasma collection — Approximately 3mL of blood will be taken from each subject just prior to the colonoscopy.
Procedure: Cervical and Vaginal Biopsy — 2 biopsies each will be collected from the vaginal wall and the cervix
Procedure: Colonoscopy with Ileal and Rectal Biopsy — 10 biopsies each will be collected from the rectum and terminal ileum from each subject during the colonoscopy.

SUMMARY:
The purpose of this research study is to find out how the drugs Truvada® (tenofovir/emtricitabine), Isentress® (raltegravir), Reyataz® (atazanavir), Sustiva® (efavirenz), and Selzentry® (maraviroc) get into the intestines and the female genital tract. All of these drugs are very effective at reducing the number of HIV viruses in the blood, however it is unknown how the drugs move around inside tissues where HIV might be hiding. This study will determine specifically where in the tissue the drug and the HIV are located through the use of a new technology that takes creates a picture of the tissue. This information will help scientists determine the best way to make new drugs to target the hidden HIV in tissue.

DETAILED DESCRIPTION:
Study Design

This is an observational study of TFV, FTC, RAL, ATZ, EFV, and MVC localization within GALT (terminal ileum & rectum), vaginal, and cervical tissues in the setting of undetectable plasma HIV. Participants will be selected on the basis of receiving either TFV/FTC/RAL, TFV/FTC/ATZ/r, TFV/FTC/EFV, or TFV/FTC/MVC as part of their ongoing HIV care. After participant education, informed consent, and screening for study eligibility, participants will be evaluated at baseline. All samples will be collected over the course of a 36 hour inpatient visit as described below.

Study Sampling

1. Blood plasma will be collected after enrollment (approximately 2 hours after the start of the inpatient visit) and before the start of bowel preparation (approximately 2-12 hours after the start of the inpatient visit).
2. Vaginal and cervical tissue will be collected after enrollment (approximately 2 hours after the start of the inpatient visit) and before the start of bowel preparation (approximately 2-12 hours after the start of the inpatient visit).
3. Rectal and terminal ileal tissue will be collected at approximately 18 hours after the initiation of the bowel preparation.

Pharmacokinetic Analysis All blood, cervical, vaginal, ileal and rectal tissue samples will be analyzed by the Clinical Pharmacology and Analytical Chemistry Laboratory (CPAC) at the UNC School of Pharmacy, which is directed by the principal investigator, Angela Kashuba, PharmD. To visualize ARV localization within a tissue, one biopsy from each tissue site will be analyzed by IR-MALDESI using a previously established workflow for our laboratory.

HIV localization within tissues will be performed using in situ hybridization (ISH) in collaboration with the Haase lab at the University of Minnesota. This group has substantial experience in HIV RNA detection from human tissues, and preliminary studies have confirmed our ability to detect HIV RNA from serial slices of tissues.

Localization within tissue slices will be evaluated by IR-MALDESI. Measurement of the distribution of each ARV within pre-specified anatomical sub-regions across a tissue slice will allow for identification of areas where drug is either concentrating or lacking. ISH and IHC analysis of serial tissue slices will allow us to co-localize ARVs with HIV and HIV target cells. Once these anatomical areas have been visually identified, imaging software will be used to isolate and quantify the signal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy HIV-positive female subjects between the ages of 18 and 65 years, inclusive on the date of screening, with an intact gastrointestinal tract, uterus, and cervix. Healthy is defined as no clinically relevant abnormalities that would interfere with the interpretation of results, or pose unnecessary risk onto volunteers due to study procedures.
2. All subjects must have an undetectable viral load at the time of screening or a documented undetectable viral load within the preceding 3 months of screening.
3. All subjects must be receiving one of the study regimens as part of their regular HIV care for at least 6 months preceding the date of enrollment.
4. Subjects must not have a history of GI disease (e.g. Crohn's disease, irritable bowel syndrome, ulcerative colitis, diverticulitis, colon cancer) or have a history of GI surgery.
5. All subjects (of childbearing potential) must have a negative serum pregnancy test at screening and negative urine pregnancy tests on days of sampling and should be using at least one of the following methods of contraception from the screening visit through 72 hours prior to inpatient admission (at which time the women will be asked to remain abstinent until after their follow-up visit):

   1. Systemic hormonal contraceptive (oral, depot, transdermal or implant)
   2. IUD placed at least 1 month prior to study enrollment
   3. Bilateral tubal ligation (Sterilization)
   4. Vasectomized male partners
   5. Condom + Spermicide
   6. Engaged in sexual activity with female only sex partners or abstinent for at least 3 months prior with no intention of becoming sexually active during the study period. Any history of recent or present concomitant male sex partners will be addressed and ruled out in the context of screening participants for eligibility for the protocol
6. Body Mass Index (BMI) of approximately 18 to 37 kg/m2; and a total body weight > 45 kg (99 lbs).
7. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
8. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
9. Subject must have documentation of a normal pap smear within 36 months of the screening visit, no procedures for abnormal cervical/vaginal pathology in the last six months, at least one prior gynecological visit as part of subject's routine medical history.
10. Not receiving any known CYP3A4 inducers (rifampin, carbamazepine, St. John's wort) or inhibitors (ketoconazole, non-DHP calcium channel blockers, macrolide antibiotics) other than those contained in their HIV regimen for at least 6 months prior to enrollment.
11. Subject must be willing to abstain from sexual intercourse, douching, and all intravaginal and intrarectal objects and products for at least 72 hours prior to enrollment until study completion.
12. Subject must be Hepatitis B surface antigen negative as documented on screening labs (or documented in their clinical record).
13. Subject must not be actively involved in the conception process.
14. Subject must be able to swallow pills and have no allergies to any component of the study products (i.e. bowel preparation regimen)

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including documented drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Subjects with a history of hysterectomy or cervical resection that would preclude obtaining a cervical biopsy.
3. Subjects who are pregnant, possibly pregnant or lactating.
4. Subjects with a presence of abnormal vaginal discharge bleeding at screening.
5. History of febrile illness within five days prior to enrollment.
6. A positive urine drug screen for illicit substances (e.g. cocaine, methamphetamines) that would increase risk associated with sedation.
7. Active Hepatitis B infection
8. An untreated-positive test for syphilis, gonorrhea, Chlamydia, or trichomonas at screening. Tests for these STIs will be performed on samples from both the vaginal and rectal orifices.
9. Any clinically significant laboratory chemistry or hematology result Grade 3 or greater according to the DAIDS Laboratory Grading Tables
10. Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
11. History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week.
12. Participation in a clinical trial involving genital tract or rectal biopsies within 6 months preceding enrollment.
13. Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
14. History of sensitivity to heparin or heparin-induced thrombocytopenia.
15. Allergy to lidocaine or Monsel's solution.
16. Allergy to latex.
17. Abnormal pap smear in the past 36 months
18. Any degree of ectopy or abnormality evident during the pelvic exam at screening.
19. Any condition which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the bowel preparation appropriately.
20. Unwilling or unable to comply with the dietary and concomitant drug restrictions in regard to study drug administration as outlined in the study procedures and prohibited medications sections.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of 22 HIV positive women between 18-65 years of age (inclusive) with an intact gastrointestinal tract, uterus and cervix who are available to complete all study procedures at UNC.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Antiretroviral tissue localization | Samples collected within 24 hours post-dose
  Tissues collected during inpatient stay will be frozen for later analysis (i.e. MSI-derived images of TFV, FTC, RAL, ATZ, EFV, and MVC localization within tissue slices.) to be completed within 6 months of tissue collection.

SECONDARY OUTCOMES:
Quantitation of antiretroviral tissue concentrations by LC-MS/MS | Samples collected within 24 hours post-dose
  Tissues collected during inpatient stay will be frozen for later analysis (i.e. TFV, FTC, RAL, ATZ , EFV, and MVC concentrations in tissues as determined by LC-MS/MS) to be completed within 6 months of tissue collection.
Immunohistochemical images of CD3, CD4, and CD8 distribution within tissue slices | Samples collected within 24 hours post-dose
  Tissues collected during inpatient stay will be frozen for later analysis (i.e. IHC staining for localization of HIV target cells within serial slices of tissue) to be completed within 6 months of tissue collection.
in-situ hybridization images of HIV RNA distribution within tissue slices | Samples collected within 24 hours post-dose
  Tissues collected during inpatient stay will be frozen for later analysis (i.e. ISH staining for localization of HIV RNA within serial slices of tissue) to be completed within 6 months of tissue collection.
Quantification of antiretroviral tissue concentrations by MSI | Samples collected within 24 hours post-dose
  Tissues collected during inpatient stay will be frozen for later analysis (i.e. TFV, FTC, RAL, ATZ , EFV, and MVC concentrations in tissues as determined by MSI) to be completed within 6 months of tissue collection.

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson CG, Bokhart MT, Sykes C, Adamson L, Fedoriw Y, Luciw PA, Muddiman DC, Kashuba AD, Rosen EP. Mass spectrometry imaging reveals heterogeneous efavirenz distribution within putative HIV reservoirs. Antimicrob Agents Chemother. 2015 May;59(5):2944-8. doi: 10.1128/AAC.04952-14. Epub 2015 Mar 2. PMID 25733502
- [Background] Robichaud G, Garrard KP, Barry JA, Muddiman DC. MSiReader: an open-source interface to view and analyze high resolving power MS imaging files on Matlab platform. J Am Soc Mass Spectrom. 2013 May;24(5):718-21. doi: 10.1007/s13361-013-0607-z. Epub 2013 Mar 28. PMID 23536269